CLINICAL TRIAL: NCT05684913
Title: Cukurova University Faculty of Dentistry
Brief Title: The Effects of Zn-containing Granulate on Patient Morbidity and Wound Healing After Free Gingival Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Mustafa Ozcan, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CukurovaU-4
Record Dates: First submitted 2022-12-14; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Surgery
Keywords: free gingival graft surgery; surgical stent; zinc; pain; bleeding
MeSH Terms: conditions — Pain; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator assessing the clinical outcomes is blinded to the study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc granulate group (Experimental): The patients in this group will receive a chair-side prepared surgical stent from Zn granulates on the palatal wound after FGG surgery.
  Interventions: Procedure: Zn granulate stent after FGG surgery
- Hemostatic agent group (Active Comparator): The patients in this group will receive hemostatic agent sutured on the palatal wound after FGG surgery.
  Interventions: Procedure: Hemostatic agent suturing

INTERVENTIONS:
Procedure: Zn granulate stent after FGG surgery — Immediately after FGG harvesting from the palatal tissue, homeostasis was achieved by sterile wet gauzes and the ZnG was prepared according to the manufacturer guidelines. Briefly, approximately 10 grams of granulate was poured into hot water and then manually shaped to cover the surgical area. The retention was achieved from the palatal, occlusal and buccal surfaces of the teeth. The patient was asked to wear the ZnG for 7 days except for eating.(
  Arms: Zinc granulate group
Procedure: Hemostatic agent suturing — Immediately after FGG harvesting from the palatal tissue, homeostasis was achieved by sterile wet gauzes. Then hemostatic agent containing cellulose were sutured on the palatal wound area with 4.0 vicryl sutures in this group. Sutures were removed after 7 days.
  Arms: Hemostatic agent group

SUMMARY:
There is no study in the literature showing the effects of Zn on wound healing after free gingival graft (FGG) operation. The aim of this randomized clinical study was to compare the early healing results of the palatal wound after FGG harvesting by sterile hemostatic agent suturing or the use of surgical stent from thermoplastic Zn-containing granules which was prepared chairside.

DETAILED DESCRIPTION:
There are many studies reporting paresthesia, herpetic lesion, mucocele, excessive bleeding and severe postoperative pain after procedure.The highest pain level perceived in the palatal region after the FGG operation is experienced on the first day after the operation and decreases to the preoperative levels approximately 2 weeks after the operation. Although hemostatics, bioactive substances, antibacterial and antiseptic agents, herbal effective products, platelet concentrations, low-dose laser applications, palatal stents are used in the palatal region to accelerate the healing stages and prevent such complications, an ideal support has not been found.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal and systemically healthy

  * ≥19 years old
  * Amount of attached gingival width in the maxillary or mandibular anterior region <2 mm
  * Full mouth plaque index score, bleeding index score on full-mouth probing <15%

Exclusion criteria;

* Previously undergone surgery for a graft harvested from the palate
* Presence of systemic disease
* Taking medication known to interfere with periodontal health
* Smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | post operative 8 weeks
  Pain was scored from 0 to 10 experienced by the patients as a result of palatal wound (0: no pain, 1: minimal pain, 10: severe pain).

SECONDARY OUTCOMES:
Bleeding | post operative 7 days
  Bleeding of the palatal wound was described as prolonged hemorrhaging after the surgery and was recorded 'yes' or 'no'
Burning sensation | post operative 8 weeks
  BS was assessed as the level of sense of burning of the palatal wound via Visual Analogue Scale (0:absent 10:severe burning)
Change in dietary habits | post operative 8 weeks
  evaluated according to inability to chew resulting from the presence of the palatal wound via Visual Analogue Scale (0: no changes 10: not capable of eating)
Complete epithelization | post-operative 8 weeks
  evaluated clinically with the 3% Hydrogen Peroxide test. While the H2O2 epithelial barrier is intact, it doesn't diffuse into the connective tissue, and oxygen isn't released. The absence of bubbles after H2O2 application was considered as CE positive, and CE was recorded as a triple variable
Patient discomfort | post-operative 8 weeks
  PD was assessed by application of air spray for 5 seconds over the palatal site and then patients scored the VAS considering sensitive function (0: no discomfort, 10: extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Cenk Haytac, Study Director — Professor
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No